CLINICAL TRIAL: NCT06236321
Title: Analysing if Chemoradiotherapy Treatment in Rectal Cancer Can be Predicted by Fast Field Cycling Imaging and Microbiota Sampling. The Microbrect-FFC Study
Brief Title: The Microbrect-FFC Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2-101-21
Record Dates: First submitted 2023-08-30; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rectal cancer patients (Experimental): Patients with locally advanced rectal cancer who require neoadjuvant chemoradiotherapy
  Interventions: Other: Fast Field Cycling MRI scan; Other: Provision of saliva and faecal samples

INTERVENTIONS:
Other: Fast Field Cycling MRI scan — Three scans to be done over the period of cancer treatment
Other: Provision of saliva and faecal samples — Three times over the period of cancer treatment

SUMMARY:
This study will focus on two points:

1. To determine if response to neoadjuvant chemoradiotherapy treatment in rectal cancer can be predicted by analysing data from Fast Field Cycling imaging (FFC), a novel type of MRI technique.
2. To determine if there is evidence that the bacteria living in our mouth and in our large bowel influence the way our body responds to cancer treatment.

Rectal cancer which is locally advanced is often managed with pre-operative chemoradiotherapy. The idea is to reduce the size of the cancer and increase the chance of a complete resection at the time of an operation. Interestingly, in approximately 20% of patients a complete response (with no evidence of residual tumour) occurs. As yet, there is no mechanism to predict for complete response before treatment. In this study we seek to assess whether FFC or the microbiota can correlate with response.

In this study 60 patients with rectal cancer requiring chemoradiotherapy before surgery will be asked to take part. Each patient will have up to three FFC scans. One scan will be done prior to commencement of neoadjuvant chemoradiotherapy, the second will be arranged for seven to eight weeks after the patient has completed the preoperative treatment and the third will be done before any subsequent surgery (if required). Participants will also be asked to give saliva and bowel motions samples before chemoradiotherapy, and after eight weeks. These samples will have the type and number of bacteria analysed, as well as levels of key products of these bacteria.

The FFC imaging scans and the microbiota of the saliva and faecal samples will be analysed and results compared to the response to chemoradiotherapy using standard criteria agreed upon at the regional colorectal cancer Multidisciplinary clinical team meeting.

DETAILED DESCRIPTION:
Sixty patients with locally advanced rectal cancer who require neoadjuvant chemoradiotherapy will be included. Patients will be identified at the Colorectal Cancer (CRC) Multidisciplinary Team (MDT) meeting when a diagnosis of rectal cancer is made. Patients will then meet the consultant to confirm the standard plan for treatment.

An out-patient appointment will be arranged for the patient to see a clinical oncologist. At this appointment the rationale, practical aspects and potential side effects of pre-operative therapy will be discussed. At this point the consultant will make the patient aware of the study. A written patient information sheet will be given to the patient to consider at home. Patients will be asked to contact a member of the team if they wish to take part.

If the participant agrees to take part written informed consent will obtained at their next hospital visit. Emphasis will be made to the patient that this study will not change the clinical management of their cancer. Pelvic radiotherapy is given as an out-patient. The first step is contouring the relevant anatomy, including tumour and associated lymph nodes, as well as normal organs that we want to limit the dose of radiation received. This contouring and preparation of a radiotherapy plan (for VMAT) can take up to two weeks so there is plenty of time for the first FFC scan and sampling to be done before treatment commences.

For patients who decide to enter the study, their first FFC imaging scan will be performed before starting the pelvic radiotherapy as an out-patient. The FFC imaging scans will take place in the PEDRI unit of the Biomedical Physics Building, Foresterhill, Aberdeen. All participants will complete an MRI safety screening form before having the scan. As for conventional clinical MRI scans, time and privacy will be given for the participants to change clothes and a safe will be provided to store their valuables during the scan. The scanning procedure will be explained to them before the scan, and they will be in audio contact with the scan controller for the duration of the scan. An alarm bell will be provided for them to signal any problems. The scan will be interrupted any time that a participant asks, and they will be able to stop the procedure and leave whenever they want to, without being asked for a reason.

The FFC imaging procedure will take up to 60 minutes and will include calibrations, navigator images and a T1 dispersion sequence, which will measure the T1 maps between 200 millitesla and 20 microtesla. After the scan, the participants will be given privacy to get dressed and will have access to the safe to collect their belongings. This scan will not delay the start of their clinical therapy and will occur in the two-week gap of radiotherapy planning required by the oncology team.

The oral sample will be collected in the radiotherapy department prior to the first NaT treatment, and the patient can choose to collect the faecal sample either at home or in the clinic, both on the day they are due to start the chemoradiotherapy. Sample kits will be provided to those who wish to collect their sample at home.

On the next visit, the patient will receive treatment as normal. On completion there will be a 7 to 8 week wait to allow the treatment to have an effect on the tumour, as well as allowing for any side effects to settle. After this gap, the patient will have their second FFC scan and will be asked to provide their second faecal and saliva sample. They will also have a pelvic MRI scan which will be reviewed at the Multi-Disciplinary Team, to assess if operation planes are now clear, allowing the patient to proceed to potentially curative surgery. Patients with a clear CRM will be asked to undertake their last FFC scan prior to surgery. During surgery a specimen will be collected from theatre and brought directly to the pathology department as per standard practice. The tumour itself will be assessed using a standardised approach, and any response graded using a validated and published system 6, 13. Patients who do not undergo surgery will be assumed to have a complete response and placed in this group for analysis

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18 and above
* Patients with locally invasive rectal adenocarcinoma cancer clinically requiring neoadjuvant chemoradiotherapy
* Participants who meet the safety criteria for undergoing an MRI scan.
* Participants who can pass through a 50 cm-diameter circular hoop to ensure they will be able to fit inside the scanner
* Participants must be able to give fully informed consent.
* Participants must be mobile enough to be positioned onto the FFC scanner couch.
* Patients willing to provide faecal and saliva samples on two occasions

Exclusion Criteria:

* MRI-incompatible conditions, as detected in the MRI safety screening sheet
* Patients with early rectal cancers
* Patients with squamous cell cancers
* Patients with colon cancers
* Patients presenting as an emergency with an obstructing rectal cancer
* Patients who are treated with short course radiotherapy alone rather than long course chemoradiotherapy
* Participants under 18 years old.
* Participants who are unable to communicate in English.
* Participants who are unable to give fully informed consent.
* Women who are pregnant.
* Restrictions to mobility that would prevent the correct positioning in the scanner.
* Patients who suffer from claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
To assess if subsets of Rectal Cancers can be correlated with FFC scan hydrogen ion dissociation curves | 12 months
  We will analyse hydrogen ion relaxation curves and correlate these curves with response to neoadjuvant chemoradiotherapy. Response has been standardised into Complete, Good partial, partial and minimal and these have been validated in previous studies. We will assess whether changes in hydrogen ion relaxation curves between rectal cancer patients can link with these response categories.

SECONDARY OUTCOMES:
To determine acceptability of FFC imaging to patients with rectal cancer by analysing patient feedback | 12 months
  Completion of feedback questionnaire
To determine correlation between faecal microbial composition and response to neoadjuvant chemoradiotherapy | 12 months
  We will undertake 16srRNA pyrosequencing of faecal samples from the patients who are having these FFC scans and correlate these analysis with reponse to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided